CLINICAL TRIAL: NCT02907970
Title: Identification Des barrières au dépistage du Cancer du Col utérin à la Réunion et Des Leviers d'amélioration
Brief Title: Perceived Barriers of Cervical Cancer Screening in Reunion Island and Key Levers for Improvment
Acronym: FOSFORE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/CHU/FOSFORE
Record Dates: First submitted 2016-09-09; First posted 2016-09-20 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Cervical cancer; Screening; Barriers
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
FOSFORE study aims at identifying the barriers of cervical cancer screening in Reunion Island and key levers for improvment.

DETAILED DESCRIPTION:
FOSFORE is a cross sectional KABP (Knowledge, Attitudes, Beliefs and Practices) telephone survey on cervical cancer screening from a sounding board of women aged between 25 and 65 years and living in Reunion Island.

Sample size was estimated from local datas on cervical cancer screening.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 25 and 65 yo
* living in Reunion Island
* speaking French, Creole or Shimaore language
* able to answer phone

Exclusion Criteria:

* history of hysterectomy
* history of incomplete or total conisation

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Telephone survey from a sounding board of women living in Reunion Island
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Type of barriers in cervical cancer screening | 6 months
  Telephone survey with a KABP-like questionnaire
Proportion of barriers in cervical cancer screening | 6 months
  Telephone survey with a KABP-like questionnaire

SECONDARY OUTCOMES:
Type of levers in cervical cancer screening | 6 months
  Telephone survey with a KABP-like questionnaire
Proportion of levers in cervical cancer screening | 6 months
  Telephone survey with a KABP-like questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Universitaire de La Réunion, Saint-Pierre, France